CLINICAL TRIAL: NCT02600962
Title: Impact of Initial Diagnosis on Mortality for Patients Hospitalised With Acute Myocardial Infarction: A National Cohort Study
Brief Title: Impact of Initial Diagnosis on Mortality for Patients Hospitalised With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Dr Christopher Gale, Associate professor, University of Leeds
Other Study IDs: Initial diagnosis study; PG/13/81/30474 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: ST-elevation Myocardial Infarction; Non ST-elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI: Patients discharged with STEMI
- NSTEMI: Patients discharged with NSTEMI

SUMMARY:
The aim of the study is to investigate the impact of an initial non-specific / non-cardiac diagnosis on mortality among patients hospitalised with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 100 years
* patients discharged alive with STEMI or NSTEMI

Exclusion Criteria:

* patients who die in hospital
* patients not discharged with STEMI or NSTEMI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises 725,860 patients hospitalised for acute myocardial infarction and entered into the Myocardial Ischaemia National Audit Project (MINAP) database between April 2004 and March 2013.
Sampling Method: Non-Probability Sample
Enrollment: 564412 (Actual)
Dates: Start 2003-01; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Mortality | Mortality censored 1 year after discharged from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Gale, PhD, Principal Investigator — University of Leeds